CLINICAL TRIAL: NCT01563328
Title: A Phase I, Open Label, Randomized, Two Cohort, Two Period, Oneway Study to Evaluate the Effect of Boceprevir and Telaprevir onDolutegravir Pharmacokinetics in Healthy Adult Subjects (ING115697)
Brief Title: A Study to Evaluate the Effect of Boceprevir and Telaprevir on Dolutegravir Pharmacokinetics in Healthy Adult Subjects (ING115697).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Shionogi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 115697
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: Dolutegravir, GSK1349572, DTG, BCV, TVR, drug interaction
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — dolutegravir; N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; telaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): DTG x 5 days followed by BCV + DTG x 10 days
  Interventions: Drug: DTG; Drug: BCV
- Cohort 2 (Experimental): DTG x 5 days followed by TVR + DTG x 10 days
  Interventions: Drug: DTG; Drug: TVR

INTERVENTIONS:
Drug: DTG — 50 mg q24h
  Other Names: Dolutegravir
Drug: BCV — 800 mg q8h
  Other Names: Boceprevir
  Arms: Cohort 1
Drug: TVR — 750 mg q8h
  Other Names: Telaprevir
  Arms: Cohort 2

SUMMARY:
Dolutegravir (DTG, GSK1349572) is an integrase inhibitor that is currently in Phase 3 clinical development for the treatment of human immunodeficiency virus (HIV) infection. Co-infection with Hepatitis C (HCV) is common in HIV-infected subjects therefore it is expected that DTG will be coadministered with treatments for HCV. Boceprevir (BCV) and Telaprevir (TVR) are protease inhibitors for the treatment of HCV that were recently approved by the Food and Drug Administration/European Medicines Agency (FDA/EMA) and have rapidly been adopted to "standard of care" in combination with pegylated interferon and ribavarin. This is a single-center, open-label, two-cohort, two-period, one-way, study in healthy adult subjects. A total of approximately 32 subjects will be enrolled, in order to obtain 24 evaluable subjects (12 per cohort). In the first treatment period, all subjects will receive DTG 50 mg once daily for 5 days (treatment A). In period 2, subjects will receive DTG 50 mg once daily plus either BCV 800 mg q8h (treatment B) for 10 days or TVR 750 mg q8h (treatment C) for 10 days. There will be no washout between treatments. Safety evaluations and serial PK samples will be collected during each treatment period.

Subjects will have a screening visit within 30 days prior to the first dose of study drug, two treatment periods, and a follow-up visit 7-14 days after the last dose of study drug.

This study will be conducted at one center in the US, with healthy adult male and female subjects.

ELIGIBILITY:
Inclusion Criteria:

* ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). A single repeat is allowed for eligibility determination.
* Single QTcB <or= 450 msec. A single repeat is allowed for eligibility determination.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and ECG. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator agrees that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Subjects with haemoglobin, WBC or neutrophil count values outside the normal range should always be excluded from enrollment. A single repeat is allowed for eligibility determination.
* Male or female between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (<147 pmol/L) is confirmatory]. Child-bearing potential and is abstinent1 or agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until the follow-up visit.
* Body weight ≥ 50 kg for males and 45 kg for females and BMI within the range 18.5- 31.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as:

an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.

* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever islonger) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* If heparin is used during PK sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
* Unable to refrain from consumption of seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices containing these products from 7 days prior to the first dose of study medication.
* The subject's systolic blood pressure at screening visit is outside the range of 90- 140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects. A single repeat is allowed for eligibility determination.
* Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination): Males Females Heart rate <45 and >100 bpm <50 and >100 bpm PR Interval <120 and >220 msec QRS duration <70 and >120 msec QTc interval (Bazett) >450 msec

  * Evidence of previous myocardial infarction (Does not include ST segment changes associated with repolarization).
  * Any clinically significant arrhythmia, any clinically significant conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree or higher], Wolf Parkinson White [WPW] syndrome), sinus pauses>3 seconds, and non-sustained or sustained ventricular tachycardia (≥3 consecutive ventricular ectopic beats).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-03-01; Primary Completion 2012-05-01 (Actual); Study Completion 2012-05-01 (Actual)

PRIMARY OUTCOMES:
Plasma steady-state DTG PK parameters AUC(0-τ), Cmax, Cmin, and Cτ | For 24 hours after dosing on Period 1 Day 5 and Period 2 Day 10
  Samples will be collected at predose and at 1, 2, 3, 4, 6, 8, 12 and 24 hours post dose

SECONDARY OUTCOMES:
Safety and tolerability parameters as assessed by change from baseline in vital signs n(BP and HR), number of subjects with adverse events and toxicity grading of clinical laboratory tests. | Up to 29 days
Plasma steady-state DTG tmax and t1/2 | For 24 hours after dosing on Period 1 Day 5 and Period 2 Day 10
  Samples will be collected at predose and at 1, 2, 3, 4, 6, 8, 12 and 24 hours post dose
Plasma steady-state TVR and BCV AUC(0-t), Cmax, Cmin, and Ct | For 8 hours after dosing on Period 2, Day 10
  Samples will be collected at predose and at 1, 2, 3, 4, and 8 hours post dose
Plasma steady-state TVR and BCV tmax and t1/2 | For 8 hours after dosing on Period 2, Day 10
  Samples will be collected at predose and at 1, 2, 3, 4, and 8 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

REFERENCES:
- [Background] Johnson M, Borland J, Chen S, et al. The effect of boceprevir and telaprevir on dolutegravir pharmacokinetics in healthy adult subjects. Published at: International Workshop on Clinical Pharmacology of HIV Therapy - 14th Annual; April 22-24, 2013; Amsterdam, the Netherlands.
- [Derived] Johnson M, Borland J, Chen S, Savina P, Wynne B, Piscitelli S. Effects of boceprevir and telaprevir on the pharmacokinetics of dolutegravir. Br J Clin Pharmacol. 2014 Nov;78(5):1043-9. doi: 10.1111/bcp.12428. PMID 24838177